CLINICAL TRIAL: NCT06496763
Title: Assessment of an Automated Optical Coherence Tomography and Camera : Effectiveness o
Brief Title: Assessment of an Automated Optical Coherence Tomography and Camera : Effectiveness of Vision-700
Status: Completed | Type: Observational
Sponsor: Crystalvue Medical Coporation (Industry)
Responsible Party: Sponsor
Other Study IDs: Effectiveness of Vision-700
Record Dates: First submitted 2024-07-04; First posted 2024-07-11 (Actual); Last update posted 2024-07-11 (Actual); Status verified 2024-07

CONDITIONS: Normal Subject; Glaucoma; Retinal Disease; Cornea
MeSH Terms: conditions — Glaucoma; Retinal Diseases; Corneal Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Normal Group:: (1)Subjects presenting at the site with normal eyes bilaterally (cataracts are acceptable). (2)IOP ≤ 21 mmHg bilaterally; BCVA 20/40 or better bilaterally. (3) No history of corneal, glaucoma, or retinal diseases. (4)No history of ocular surgeries, including laser refractive surgery, cataract surgery, glaucoma surgery and retinal surgery. (5)Subjects without any current ocular pathology other than cataract in the normal eye(s), as determined by self-report and/or investigator assessment at the study visit.
  Interventions: Device: Vision-700
- Glaucoma Group: (1) With a current BCVA of 20/40 or better in the glaucoma study eyes. (2) History of visual field defects within the previous six months from the study visit or measured on the day of the study visit that is consistent with glaucomatous optic nerve damage. (3) Subjects who have been diagnosed with glaucoma in the glaucoma study eyes based on the presence of visual field defects, regardless of the optic nerve head and RNFL appearance. (4) Subjects without retinal disease or cornea condition in the glaucoma study eyes, as determined by self-report and/or investigator assessment at the study visit.
  Interventions: Device: Vision-700
- Retinal Disease Group: (1)Subjects with a current BCVA of 20/400 or better in the retinal disease study eye(s) at the study visit. (2)Subjects diagnosed with retinal pathology including but not limited to any one of following criteria: a. Non Exudative Macular Degeneration (dry AMD), Diabetic Macular Edema, Macular Hole, Epiretinal Membrane, Cystoid Macular Edema, or other retinal disease in the study eye(s) as confirmed within the past six months, who exhibit structural lesions in the study eye; b. Neovascular Macular Degeneration (wet AMD), Diabetic Retinopathy, Retinal Artery Occlusion, Retinal Vein Occlusion or other retinal disease in the study eye(s) as confirmed within the past six months, who exhibit vascular and/or ischemic lesions in the study eye. (3) Subjects without glaucoma or cornea condition in the retinal disease study eye(s), as determined by self-report and/or investigator assessment at the study visit.
  Interventions: Device: Vision-700
- Cornea Condition Group: History of refractive surgery, contact lens (wear contact lens more than 6 months), dry eye or keratoconus.
  Interventions: Device: Vision-700

INTERVENTIONS:
Device: Vision-700 — OCT machines used for diagnostic purposes
  Other Names: 3D OCT-1 Maestro

SUMMARY:
The objective of study is to assess the repeatability and agreement of the retina and cornea measurement by Vision-700 in comparison with those by 3D OCT-1.

DETAILED DESCRIPTION:
The first objective of study is to assess the repeatability and agreement of the retina and cornea measurement by Vision-700 in comparison with those by 3D OCT-1, and Cornea Measurements by RTVue XR + CAM. The second objective is to compare the agreement of fundus photography quality between Vision-700 with 3D OCT-1.

ELIGIBILITY:
Inclusion Criteria:

Subject 22 years old or older on the date of informed consent; Subjects able to understand the written informed consent and willing to participate as evidenced by signing the informed consent.

Normal Group:

(1)Subjects presenting at the site with normal eyes bilaterally (cataracts are acceptable). (2)IOP ≤ 21 mmHg bilaterally; BCVA 20/40 or better bilaterally. (3) No history of corneal, glaucoma, or retinal diseases. (4)No history of ocular surgeries, including laser refractive surgery, cataract surgery, glaucoma surgery and retinal surgery. (5)Subjects without any current ocular pathology other than cataract in the normal eye(s), as determined by self-report and/or investigator assessment at the study visit.

Glaucoma Group:

(1) With a current BCVA of 20/40 or better in the glaucoma study eyes. (2) History of visual field defects within the previous six months from the study visit or measured on the day of the study visit that is consistent with glaucomatous optic nerve damage. (3) Subjects who have been diagnosed with glaucoma in the glaucoma study eyes based on the presence of visual field defects, regardless of the optic nerve head and RNFL appearance. (4) Subjects without retinal disease or cornea condition in the glaucoma study eyes, as determined by self-report and/or investigator assessment at the study visit.

Retinal Disease Group:

(1)Subjects with a current BCVA of 20/400 or better in the retinal disease study eye(s) at the study visit. (2)Subjects diagnosed with retinal pathology including but not limited to any one of following criteria: a. Non Exudative Macular Degeneration (dry AMD), Diabetic Macular Edema, Macular Hole, Epiretinal Membrane, Cystoid Macular Edema, or other retinal disease in the study eye(s) as confirmed within the past six months, who exhibit structural lesions in the study eye; b. Neovascular Macular Degeneration (wet AMD), Diabetic Retinopathy, Retinal Artery Occlusion, Retinal Vein Occlusion or other retinal disease in the study eye(s) as confirmed within the past six months, who exhibit vascular and/or ischemic lesions in the study eye. (3) Subjects without glaucoma or cornea condition in the retinal disease study eye(s), as determined by self-report and/or investigator assessment at the study visit.

Cornea Condition Group:

History of refractive surgery, contact lens (wear contact lens more than 6 months), dry eye or keratoconus.

Exclusion Criteria:

1. Subjects unable to tolerate ophthalmic imaging;
2. Subjects with ocular media not sufficiently clear to obtain acceptable OCT images;
3. Subjects with a history of leukemia, dementia or multiple sclerosis.
4. Subjects with history of hydroxychloroquine or chloroquine use
5. Subjects with photosensitivity
6. Subject having Photodynamic therapy (PDT) within 6 months
7. Subjects taking photosensitivity drug currently
8. Subject has a condition or is in a situation which the investigator feels may put the subject at significant risk, may confound the study results, or may interfere significantly with the subject's participation in the study.

Min Age: 22 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Healthy subjects, Glaucoma subjects, Retinal diseasse subjects, Cornea condition subjects
Sampling Method: Non-Probability Sample
Enrollment: 159 (Actual)
Dates: Start 2022-09-01 (Actual); Primary Completion 2022-09-01 (Actual); Study Completion 2023-07-31 (Actual)

PRIMARY OUTCOMES:
The Precision of Vision-700 in Retinal and Cornea Measurement | 2022/9/1
  The Precision included the repeatability and reproducibility.
The Precision of 3D OCT-1 in Retinal and Cornea Measurements | 2022/9/1
  The Precision included the repeatability and reproducibility.
The Agreement of Vision-700 and 3D OCT-1 in Retinal and Cornea Measurements | 2022/9/1
  the agreement study

CONTACTS AND LOCATIONS:
Overall Officials: I-Chia Liang, Principal Investigator — Tri-Services General Hospital
Locations (1):
- Tri-Services General Hospital, Taipei County, Taiwan

IPD SHARING:
Plan to Share IPD: Undecided